CLINICAL TRIAL: NCT06817980
Title: Disorders of the Sense of Self and Physical Activity
Acronym: sensdesoi
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 9530
Record Dates: First submitted 2024-12-16; First posted 2025-02-10 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: SCHIZOPHRENIA 1 (Disorder); Borderline Personality Disorder; Vestibular Syndromes
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self and physical activity protocol (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — - Physical activity: We will compare the impact of 3 different environments (with no object in the environment, vs. with some objects but no hidden objects vs. with objects at the fore- and background) during (total of 9 sessions of 30 minutes + 3*5 minutes of testing), on the measure of self (see below).
  Visit 10: We will repeat a walking session. Participants will wear mixed-reality goggles, which allow them to visualize the environment and superimpose a continuous stream of light. This session is intended to test the idea that this flow would enable SZ patients to suffer less from the discontinuous appearance of information when moving around.
  Measure of 'self' : the participants will decide whether the line presented on a computer screen is static or moving. They will be immobile, walking on the spot in front of the computer, or passively mobilized with a whole-body movement platform. The latter condition will be used only in the first phase of the protocol

SUMMARY:
Schizophrenia (SZ) patients with metabolic syndrome, patients with vestibular syndrome, and patients with borderline personality disorder, would benefit from physical activity (PA). Yet patient adherence to PA is low, at least in the case of SZ. the investigators work and the literature lead the investigators to consider that, in addition to motivational aspects, disorders of the bodily sense of self could play a role in this lack of adherence. Simply walking involves visual movements related to the self, which must be distinguished from movements in the environment. This means a distinction between self and not-self. Furthermore, these movements are all the more difficult to distinguish as they may also result from the fact that hidden objects become visible as a result of our own movement. In all sense-of-self disorders can themselves affect physical training, and the investigators will measure them in the first stage. In the second stage, the investigators will apply a standard, risk-free PA protocol by walking (3x3 sessions of 30 min). the investigators will test the impact of physical training on the sense of self under different conditions, with one environment minimizing self-related movement, vs. 2 environments with a variable level of enrichment (i.e. hidden objects inducing more or less self-related movement).

At the end of the protocol, the investigators will offer participants who wish to take part in an ancillary study, i.e. a walking session with mixed-reality goggles. These will superimpose a luminous flux on the periphery of the visual field. According to results obtained in the laboratory, this flux could restore sensory mechanisms impaired in schizophrenia. the investigators will use these glasses in the most difficult condition for the patient, and verify their impact.

ELIGIBILITY:
Inclusion Criteria:

* Criteria common to all participants:
* Men or women aged 18 to 60 inclusive
* Subject affiliated to a health insurance scheme, beneficiary or beneficiary's beneficiary
* Able to understand the aims and risks of the research, and to give informed consent
* Visual acuity > 0.7 on the Freiburg Vision Test (Bach 1996) due to the use of visual equipment
* BMI (body mass index) < 40 (due to cardiovascular risk).

Patient-specific criteria:

* With schizophrenia: criteria for schizophrenia as defined in the DSMV (American Psychiatric Association, 2015)
* With borderline personality disorder: criteria for borderline personality disorder as defined in the DSMV (American Psychiatric Association, 2015)
* With vestibular disorders: peripheral vestibular disorders established after otolaryngological examination

Exclusion Criteria:

* Criteria common to all participants:
* Serious or unstabilized somatic pathology (including cardiovascular)
* History likely to affect cerebral anatomy or to be linked to an abnormality (neonatal suffering, neurosurgical operation, comitiality, stroke...)
* Presence of joint pain, likely to worsen after exercise
* - Substance use disorders (as defined by DSM-IV TR)
* 3D vision disorders as measured by the Wirt stereotest (depth perception at a disparity of at least 80'' arc)
* Movement perception disorders (correct movement discrimination in less than 75% of trials (cf. § V-2.2)
* History of general anaesthesia in the 3 months preceding the study
* History of neurological disease
* Impossibility of giving the subject informed information (subject in emergency situation)
* Pregnancy declared by patient
* Breast-feeding
* Subject in exclusion period (determined by a previous or current study)
* Subject hospitalized
* Subject under court protection

Exclusion criteria specific to control subjects or patients with vestibular syndrome:

History of major psychiatric pathology with current psychotropic medication (i.e., antidepressant, thymoregulator, antipsychotic)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Impact of physical activity on the 'self' measure | Day 0
  Quantification of the d' index, which represents the ability to discriminate between moving and static lines (whose movement is only related to one's own displacement, which induces a mirror movement on the retina). The d' will be measured three times per PA session, and in all 3 sessions per condition (neutral vs. enriched, with increasing complexity of self-related movements).
  The evaluation criterion will be the evolution of the d' index over the course of the PA training sessions in the 3 conditions.
Impact of physical activity on the 'self' measure | between Day 0 and Month 3
  Quantification of the d' index, which represents the ability to discriminate between moving and static lines (whose movement is only related to one's own displacement, which induces a mirror movement on the retina). The d' will be measured three times per PA session, and in all 3 sessions per condition (neutral vs. enriched, with increasing complexity of self-related movements).
  The evaluation criterion will be the evolution of the d' index over the course of the PA training sessions in the 3 conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de psychiatrie, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No